CLINICAL TRIAL: NCT04424147
Title: Efficacy and Safety of HVA Regimens as Salvage Treatment in Relapsed/Refractory (rr) Acute Myeloid Leukemia (AML)
Brief Title: Efficacy and Safety of HVA Regimens as Salvage Treatment in rrAML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Shenzhen Second People's Hospital (Other); The Seventh Affiliated Hospital of Sun Yat-sen University (Other); Maoming People's Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Shenzhen Hospital, Southern Medical University (Unknown); Shanghai Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine (Unknown); The First People's Hospital of Chenzhou (Unknown); Peking University Shenzhen Hospital (Other); Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HVA in rrAML
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Refractory Acute Myeloid Leukemia; Relapsed Acute Erythroid Leukemia; Salvage Treatment; HVA Regimen
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Erythroblastic, Acute | interventions — Salvage Therapy

STUDY DESIGN:
Intervention Model Description: Patients with rrAML are treated with HVA regimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HVA treatment (Experimental): All patients with rrAML are treated with HVA regimen
  Interventions: Combination Product: HVA Regimens as Salvage Treatment

INTERVENTIONS:
Combination Product: HVA Regimens as Salvage Treatment — venetoclax with a dose of 400mg per day for 14 days, combined with azacitidine (AZA) with a dose of 75mg/m2 per day for 7 days, and HHT 1mg/m2 per day for 7 days

SUMMARY:
Up Until now, there is not well acepted treatment for relapsed/refractory (rr) acute myeloid luekemia (AML), which has low complete response and poor survival. According to different guildlines, clinical trial is the first choice for the treatment of rrAML. High expression of BCL-2 and hypermethylation are very important factors for drug resistance in AML. Lots of studies have reported combination of BCL-2 inhibitor with hypomethylating agents (HMA) showed a promising efficacy in elder or unfit patients with newly diagnosed AML, however, presented not that exciting curing effect in rrAML. It is known that overexpression of MCL-1 and BCL-XL is the main reason for leukemia cells being resistant to BCL2 inhibitors. Since Homoharringtonine (HHT) could downregulate MCL-1 and BCL-XL in leukemia cells, there might be a synergic effect for combination of BCL-2 inhibitors with HHT, which has been proven in the treatment of lymphoma. Yet, there is not a report for the use of this combination in AML. In this single arm multi-centers prospective study, adult patients with rrAML are included and treated with BCL-2 inhibitor venetoclax at a dose of 400mg per day for 14 days, combined with azacitidine (AZA) at a dose of 75mg/m2 per day for 7 days, and HHT 1mg/m2 per day for 7 days, and then the eficacy and safety of HVA regimens as salvage treatment in rrAML are assessed.

ELIGIBILITY:
Inclusion Criteria:

Patients with rrAML Patients with the age of 18-65 years old

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Complete response | At the end of Cycle 2 (each cycle is 28 days)
  Blast rate lower than 5% with or without peripheral blood cell recover

SECONDARY OUTCOMES:
Safety and Tolerability of HVA treatment | At the end of Cycle 2 (each cycle is 28 days)
  The number of participants experiencing 3/4 degree bone marrow suppession and infection.
Disease-free survival | one year
Overall survival | one year

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu S, Zhang Y, Yu G, Wang Y, Shao R, Du X, Xu N, Lin D, Zhao W, Zhang X, Xiao J, Sun Z, Deng L, Liang X, Zhang H, Guo Z, Dai M, Shi P, Huang F, Fan Z, Liu Q, Lin R, Jiang X, Xuan L, Liu Q, Jin H. Sorafenib plus triplet therapy with venetoclax, azacitidine and homoharringtonine for refractory/relapsed acute myeloid leukemia with FLT3-ITD: A multicenter phase 2 study. J Intern Med. 2024 Feb;295(2):216-228. doi: 10.1111/joim.13738. Epub 2023 Oct 29. PMID 37899297
- [Derived] Jin H, Zhang Y, Yu S, Du X, Xu N, Shao R, Lin D, Chen Y, Xiao J, Sun Z, Deng L, Liang X, Zhang H, Guo Z, Dai M, Shi P, Huang F, Fan Z, Yin Z, Xuan L, Lin R, Jiang X, Yu G, Liu Q. Venetoclax Combined with Azacitidine and Homoharringtonine in Relapsed/Refractory AML: A Multicenter, Phase 2 Trial. J Hematol Oncol. 2023 Apr 29;16(1):42. doi: 10.1186/s13045-023-01437-1. PMID 37120593